CLINICAL TRIAL: NCT03975114
Title: A Randomized Phase 2 Study Comparing Immunotherapy With Chemotherapy in the Treatment of Elderly Patients With Advanced NSCLC (MILES-5)
Brief Title: A Study Comparing Immunotherapy With Chemotherapy in the Treatment of Elderly Patients With Advanced NSCLC (MILES-5)
Acronym: MILES-5
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: University of Campania Luigi Vanvitelli (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MILES-5
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Eldelry; metastatic Non-Small-Cell Lung Cancer; Durvalumab; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: Comparative Randomized Phase 2 Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Chemo first (Active Comparator): Standard chemotherapy followed at progression by durvalumab
  Interventions: Drug: Chemotherapy; Drug: Durvalumab
- Immuno Monotherapy first (Experimental): Experimental single agent immunotherapy with durvalumab followed at progression by chemotherapy
  Interventions: Drug: Chemotherapy; Drug: Durvalumab
- Immuno Combination Therapy first (Experimental): experimental single agent immunotherapy with durvalumab followed at progression by chemotherapy
  Interventions: Drug: Chemotherapy; Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Chemotherapy — Any approved first line chemotherapy regimen at Investigators' choice
Drug: Durvalumab — Durvalumab 1500 mg iv Q4w until progressive or unacceptable toxicity or patient's refusal
Drug: Tremelimumab — Tremelimumab 75 mg iv Q4w for 4 administrations (4 months)
  Arms: Immuno Combination Therapy first

SUMMARY:
This is a randomized phase 2 trial aiming to assess the early efficacy of two experimental treatment sequences.

Three arms are planned; (i) standard chemotherapy followed at progression by single agent immunotherapy with durvalumab (CT), (ii) experimental single agent immunotherapy with durvalumab followed at progression by chemotherapy, (iii) experimental combination immunotherapy with durvalumab+tremelimumab followed at progression by chemotherapy.

The the two experimental strategies will be compared with the standard strategy in terms of 12-month overall survival, time considered informative for the type of treatment and disease

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >= 70 years of age.
2. Histological documentation of primary squamous or non squamous non-small cell lung carcinoma.
3. Availability of archived tumor tissue block or newly cut unstained slides for PD-L1 determination.
4. Stage IV or IIIB disease with supraclavear metastatic nodes (according to TNM 7th edition).
5. Clinical or radiologic evidence of disease (at least one measurable or non measurable lesion).
6. ECOG performance status 0 to 1.
7. Life expectancy > 3 months.
8. Adequate renal and hepatic function, defined as:

   1. Total serum bilirubin ≤ 1.5 institutional ULN.
   2. AST and/or ALT ≤ 2.5 x ULN for the institution (or ≤ 5 x ULN if liver metastases are present)
   3. Serum creatinine ≤ 1.5 x ULN for the institution (or calculated creatinine clearance ≥ 40 mL/min/1.73 m2).
9. Adequate bone marrow function, defined as:

   1. Haemoglobin <= 9.0 g/dL
   2. Absolute neutrophils count (ANC) >= 1.5 x 109/L (> 1500 per mm3)
   3. Platelet count <= 100 x 109/L(>100,000 per mm3).
10. Written informed consent obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

Cancer related

1. Activating epidermal growth factor receptor mutation (exon19 deletion or exon 21 L858R mutation or other activating/sensitizing mutations).
2. ALK or ROS1 positive (immunohistochemistry or FISH)
3. Mixed small-cell lung cancer and NSCLC histology.

   Prior, current or planned treatment related
4. Prior chemotherapy or any other medical treatment for advanced NSCLC (previous neoadjuvant or adjuvant chemotherapy is allowed if > 6 months previously).
5. Prior exposure to immunomodulatory therapy, including, but not limited to, other anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4), anti-programmed cell death1 (PD-1), anti-programmed cell death ligand 1 (PD-L1), or anti PD-L2 antibodies.
6. Current or prior use of immunosuppressive medication within 14 days before the first dose of study treatment (intranasal and inhaled corticosteroids at physiological doses not exceeding 10 mg/day of prednisone or an equivalent corticosteroid are allowed).
7. Any concurrent investigational product or other anticancer treatment.

   Prior or concomitant conditions or procedures related
8. Active or prior documented autoimmune disease within the past 2 years (subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment within the past 2 years, are not excluded).
9. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
10. History of allogeneic organ transplant
11. History of active primary immunodeficiency.
12. Active infection, including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
13. Receipt of live attenuated vaccine within 30 days prior to the first dose of study drugs.
14. Patients with previous malignancies (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer or surgically resected prostate cancer with normal PSA) are excluded only if the histological diagnosis of the current disease does not definitely support the pulmonary origin.
15. Brain metastases or spinal cord compression, unless asymptomatic, previously treated, and stable off steroids and anti-convulsants for at least one month prior to study entry.
16. Leptomeningeal carcinomatosis
17. Clinically significant cardiovascular disease, including:

    1. Myocardial infarction or unstable angina pectoris within < 6 months prior to the first study treatment
    2. New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF)
    3. Uncontrolled hypertension
    4. Serious cardiac arrhythmia requiring medication (with the exception of atrial fibrillation or paroxysmal supraventricular tachycardia)
    5. Peripheral vascular disease > grade 3 (i.e. symptomatic and interfering with activities of daily living requiring repair or revision)
    6. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction.
18. Serious active infection requiring i.v. antibiotics at enrollment.
19. Known hypersensitivity to any of the study drugs or excipients.
20. Evidence of any other concomitant pathologies, physical examination or laboratory findings (including but not limited to active peptic ulcer disease or gastritis, active bleeding diatheses or psychiatric illness) or social situation that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment related complications.
21. Radiotherapy treatment to the chest or to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study treatment (patients who have had radiotherapy ≥ 4 weeks prior to the first dose of study treatment, but who are still experiencing acute toxic effects of radiotherapy are also excluded).
22. Major surgical procedure within 28 days prior to the first dose of study drugs.
23. Male patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of study treatment.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
12-month overall survival | 12 months
  12-month overall survival is defined as the Kaplan-Meier (K-M) survival probability at 12 months after randomization (Chen 2015).

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Perrone, MD, PhD, Study Chair — Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale
Locations (1):
- Istituto Nazionale Tumori, IRCCS, Fondazione G. Pascale, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available at request